CLINICAL TRIAL: NCT05274607
Title: French Epidemiological Pediatric Study on Pneumonia and Empyema in Emergency Departments in Children 1 Month to 15 Years
Brief Title: Pneumonia and Empyema in Emergency Departments in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: ACT0209
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Pneumonia; Pleural Effusion
Keywords: children; pneumococcal conjugate vaccine
MeSH Terms: conditions — Pneumonia; Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Describe the epidemiology of hospitalized pediatric pneumonia and pneumonia with pleural effusion: frequency, clinical and biological characteristics, responsible bacteria and pneumococcus place, antibiotic resistance, treatment, vaccine status.

DETAILED DESCRIPTION:
The pneumonia observatory began in June 2009 and has included more than 15,000 children with pneumonia or pneumonia with pleural effusion (hospitalized or not) until May 2019. This study led to the publication of many articles in international peer-reviewed journals. Since June 2019, the scientific committee of the study met at the ESPID congress has decided to include only hospitalized patients. This amendment is justified for three reasons:

* Change in criteria for diagnosing pneumonia with increasing use of chest ultrasound
* Logistical aspects and workload of investigating centers too important
* Long-term impact of pneumococcal vaccine 13-valent especially marked for the most severe cases In this context, the purpose of this amended study is to enroll only the most severe cases of pneumonia, i.e. requiring hospitalization, in ICU or not. Since this study began in 2009, we have already enrolled hospitalized cases, we will have a baseline prior to the introduction of third-generation PCVs (pneumococcal conjugate vaccines) and we will be able to continue monitoring with data since 2009.

ELIGIBILITY:
Inclusion Criteria:

* ages between 1 month and 15 years
* presence of parenchymatous condensation and/or pleural effusion on chest x-rays and/or ultrasounds and/or CT scans
* fever ≥38.5 °C if age ≥3 months since the onset of symptoms or ≥38 °C if the child is less than 3 months old.
* Hospitalization

Exclusion Criteria:

* Refusal of participation by the patient, his or her relative or legal representative (depending on the situation)

Ages: 1 Month to 15 Years | Sex: All
Age Groups: Child
Study Population: Hospitalized children presenting with pneumonia or pleural effusion
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2009-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Epidemiology of hospitalized pediatric pneumonia and pneumonia with pleural effusion | 15 years
  - Describe the epidemiology of hospitalized pediatric pneumonia and pneumonia with pleural effusion: frequency, clinical and biological characteristics, responsible bacteria and pneumococcus place, antibiotic resistance, treatment, vaccine status.

SECONDARY OUTCOMES:
Impact of pneumococcal conjugate vaccines | 15 years
  Measuring the impact of PCV vaccines on pneumonia and pleural effusion
Treatments | 15 years
  Describe the therapeutics in place

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cohen, MD, Study Director — Groupe de Pathologies Infectieuses Pédiatriques (GPIP)
Locations (1):
- ACTIV, Créteil, France